CLINICAL TRIAL: NCT04351737
Title: DEXTENZA for the Treatment of Post-Surgical Pain and Inflammation ComparEd to StandaRd of Care Topical Cortico-Steroid Treatment In PatientS Who Undergo BilaTeral Pterygium Surgery PERSIST Study
Brief Title: Dextenza for Post-operative Treatment of Pterygium
Acronym: PERSIST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brandon Eye Associates, PA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PERSIST Study
Record Dates: First submitted 2020-03-11; First posted 2020-04-17 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Pterygium of Both Eyes
MeSH Terms: interventions — Mutagenesis, Insertional; Calcium Dobesilate; prednisolone acetate

STUDY DESIGN:
Intervention Model Description: In patients who undergo bilateral pterygium surgery, eyes will be randomized to receive either DEXTENZA at baseline, Month 1 and Month 2 or prednisolone x 3 months. Both eyes will receive antibiotic drops four times per day for two weeks and Maxitrol ointment at bedtime for two weeks following surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pterygium patients (Experimental): patients with bilateral pterytium
  Interventions: Drug: Intracanalicular Dexamethasone, (0.4 mg) Insert; Drug: Prednisolone Acetate

INTERVENTIONS:
Drug: Intracanalicular Dexamethasone, (0.4 mg) Insert — To determine post-surgical resolution of pain and inflammation outcomes with DEXTENZA compared to topical steroid treatment in patients who undergo bilateral pterygium surgery.
  Other Names: Dextenza
Drug: Prednisolone Acetate — To reduce post-surgical pain and inflammation in patients who undergo bilateral pterygium surgery.

SUMMARY:
DEXTENZA for the Treatment of Post-Surgical Pain and Inflammation Compared to Standard of Care Topical Cortico-steroid Treatment in Patients who Undergo Bilateral Pterygium Surgery

DETAILED DESCRIPTION:
In patients who undergo bilateral pterygium surgery, eyes will be randomized to receive either DEXTENZA at baseline, Month 1 and Month 2 or prednisolone x 3 months. Both eyes will receive antibiotic drops four times per day for two weeks and Maxitrol ointment at bedtime for two weeks following surgery.

ELIGIBILITY:
Inclusion Criteria: patients with bilateral pterygium -

Exclusion Criteria: none

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Patient pain level follow pterygium removal | 2 months
  measurement of pain following pterygium removal using the validated "Numeric Pain Rating Scale" to assess pain, which ranges from 0 to 10 with higher values indicating more severe pain.
inflammation | 2 months
  measurement of ocular surface inflammation using the standard 1+ - 4+ rating scale commonly used in ophthalmology with 4+ indicating the most inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- Brandon Eye Associates, Brandon, Florida, United States

IPD SHARING:
Plan to Share IPD: No